CLINICAL TRIAL: NCT06966726
Title: Positive Pre-Visit Imagery Does Not Reduce Dental Anxiety in Children: A Randomized, Triple-Blind, Controlled Trial
Brief Title: Positive Pre-Visit Imagery Does Not Reduce Dental Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Lavínia Lourenço Costa, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 71431923.0.0000.5537
Record Dates: First submitted 2025-04-29; First posted 2025-05-13 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Dental Anxiety; Dental Fear and Anxiety
Keywords: dental anxiety; pediatric dentistry
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Imagery Group (Experimental): Participants were exposed to positive images related to dental care (e.g., smiling children after treatment, positive interactions with the dentist) for 2 minutes prior to the dental procedure.
  Interventions: Behavioral: Positive Dental Imagery
- Neutral imagery group (Placebo Comparator): Participants were exposed to neutral images (nature scenes) for 2 minutes prior to the dental procedure.
  Interventions: Behavioral: Neutral Nature Imagery

INTERVENTIONS:
Behavioral: Positive Dental Imagery — Children were shown four A4-sized laminated color images depicting positive dental scenes (e.g., children interacting happily with the dentist, smiling after treatment) for 2 minutes prior to the procedure.
  Arms: Positive Imagery Group
Behavioral: Neutral Nature Imagery — Children were shown four A4-sized laminated color images depicting neutral nature scenes (e.g., a beach, sunset, flowers) for 2 minutes prior to the procedure.
  Arms: Neutral imagery group

SUMMARY:
This randomized triple-blind clinical trial aims to evaluate the effectiveness of positive pre-visit imagery in managing dental anxiety (DA) in children aged 5 to 13 years. DA is a common barrier to dental treatment and is often triggered by procedures such as local anaesthesia. Participants were randomly assigned to view either positive dental images or neutral nature images before treatment. Anxiety levels were assessed before and after the procedure using the Venham Picture Test. The study hypothesizes that exposure to positive dental imagery prior to the appointment may reduce anxiety levels, promoting a more positive dental experience for pediatric patients.

DETAILED DESCRIPTION:
Dental anxiety (DA) is a significant barrier to dental care in children and is commonly associated with negative treatment experiences, particularly during procedures such as local anaesthesia. Children with DA are more likely to exhibit poor oral health outcomes and reduced quality of life. Behaviour management techniques (BMTs), such as distraction, tell-show-do, desensitization, and positive reinforcement, are routinely used in pediatric dentistry to help reduce anxiety and improve cooperation.

Among the newer BMTs, positive pre-visit imagery-where children view positive dental-related images prior to treatment-has shown promise. This technique is based on observational learning and aims to create positive associations with dental care. However, current evidence is limited and inconclusive.

This triple-blind randomized controlled trial investigates the effectiveness of positive pre-visit imagery in reducing DA in children. Sixty-nine children aged 5 to 13 years requiring local anaesthesia were randomly assigned to view either a series of positive dental images (intervention group) or neutral nature scenes (control group) prior to treatment. The intervention consisted of four A4 laminated images designed to elicit positive emotional responses related to dental care, while the control group viewed four neutral nature photographs.

Anxiety was assessed before and after the dental procedure using the Venham Picture Test (VPT), a validated tool for evaluating dental anxiety in children. The primary outcome was the change in anxiety level between pre- and post-treatment, and the data were analyzed using non-parametric statistical methods.

The study follows CONSORT guidelines and was approved by the Human Research Ethics Committee at the Federal University of Rio Grande do Norte. This trial aims to provide robust evidence regarding the effectiveness of positive pre-visit imagery as a non-pharmacological strategy for managing dental anxiety in children.

ELIGIBILITY:
Inclusion Criteria:

* children aged 5-13 years who were admitted to the Paediatric Dentistry Clinic of the Federal University of Rio Grande do Norte, and who required local anaesthesia during dental treatment

Exclusion Criteria:

* Children with intellectual disabilities, visual or hearing impairments and children requiring emergency treatment were excluded

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Anxiety Level (Venham Picture Test - VPT) | Day 1 (before and after the dental procedure)
  The primary outcome of this study is to evaluate the level of dental anxiety before and after the dental procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Norte - Departamento de odontologia, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kamel DO, Wahba NA, Talaat DM. Comparison between Positive Dental Images and Neutral Images in Managing Anticipatory Anxiety of Children. J Clin Pediatr Dent. 2017;41(2):116-119. doi: 10.17796/1053-4628-41.2.116. PMID 28288299